CLINICAL TRIAL: NCT03329872
Title: Neuro-Orthopedic Registry of the University Hospital of Toulouse
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 14 7321 03
Record Dates: First submitted 2017-08-21; First posted 2017-11-06 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Neurologic Disorder
Keywords: Neuro-Orthopedics; Register
MeSH Terms: conditions — Nervous System Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients follow-up in hospital will have data collection
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — data collection about symptoms without any specific clinical or biological intervention

SUMMARY:
Neuro-orthopedics corresponds to the evaluation and therapeutic management of the orthopedic consequences of damage to the central or peripheral nervous system. In case of neurological impairment, there may be joint, motor, sensory and cognitive impairments that limit the patient's activities. The management of these orthopedic problems falls within the specific framework of neuro-orthopedics because in the presence of neurological, problems are different and more complex than in classical orthopedics. In this context, a well-conducted evaluation is a prerequisite for appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient with a neurological condition that benefits:

* An injection of botulinum toxin in the context of spasticity : about 20 / week
* Pre or post-therapeutic clinical evaluation (botulinum toxin or surgery): approximately 10 / week
* Clinical or instrumental evaluation of the walking or upper limb (Physiological Functional Explorations): about 10 / week
* A medical and surgical multidisciplinary consultation about spasticity : about 15 / month
* A discussion during neuroorthopedic multidisciplinary consultation meeting about the patient's file and anomalies of walking: about 8 / month
* Implementation of a Baclofen pump (Neurosurgery): about 2 / month
* Functional surgery of the upper or lower limb (locomotor institute, orthopedic surgery and traumatology): about 4 / sem

Exclusion Criteria:

Patient (or the legal representative) who opposes the data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with central or peripheral nervous system disorders with orthopedic consequences.
Sampling Method: Non-Probability Sample
Enrollment: 976 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Neurologic symptoms | Each year until five years
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: David Gasq, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Midi-Pyrénées, France